

## **Consent Form**



**PAIR Study** 

NICU Saint Mary's Hospital Manchester M13 9WL Tel: 01612766331/857

| Study No | Hospital Name: Saint Mary's Hospital |
|---|---|
| <b>Formal Title:</b> PAIR (Paracetamol and Ibuprofen Research) Study: A randomised controlled trial comparing IV paracetamol with IV ibuprofen in the management of haemodynamically significant patent ductus arteriosus | |
| Name of Researcher:<br>Dr Arindam Mukherjee | Please initial each box |
| I,mother/ Do hereby give my consent for my baby to I | |
| I give my consent for the research team to a | access my baby's medical records. |
| I confirm that I have been given the participant information sheet (version 7, June 2021) which I have read and understood. I have been given an opportunity to ask my questions which have been answered. | |
| I can confirm that my baby's participation in this trial is entirely voluntary. I understand what will happen to my baby during this trial. I am aware of my rights to withdraw my baby from the trial at any time. In such an event if I chose to do so, his/her future care or legal rights will not be affected in any way. | |
| I also give my consent to publish the trial results in scientific journals and to present the data in national and international meetings and conferences provided no personal details will be made available at any stage. | |
| I understand that relevant sections of any of my baby's medical notes and data collected during the study, may be looked at by responsible individuals from regulatory authorities or from the NHS trust, where it is relevant to my baby taking part in this research. I give permission for these individuals to have access to my baby's records. | |
| I agree for the Neonatal unit to inform my GP about my baby's participation in this trial | |
| Name of Parent | Name of health professional taking consent |
| Signature | Date |
| Date | Signature |



Copy to – Parents
Case notes
Research Team